CLINICAL TRIAL: NCT05756075
Title: The Accuracy of Digital Assessment of Performance Trial (ADAPT): Walk Test Study
Brief Title: The ADAPT-study: Measuring Physical Performance Using Wearable Sensors in Parkinson's Disease and COPD (ADAPT)
Acronym: ADAPT
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NL78292.091.21
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease; COPD
Keywords: Physical activity; Physical capacity; Walking; Exercise; Wearable sensors; Locomotion; Home-based
MeSH Terms: conditions — Parkinson Disease; Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease
  Interventions: Behavioral: Aerobic exercise training
- COPD
  Interventions: Behavioral: Aerobic exercise training

INTERVENTIONS:
Behavioral: Aerobic exercise training — Participants will follow a personalized aerobic exercise training program twice a week at the physiotherapist. The intensity of the program is based on the results of the 6MWT according to the most recent guidelines for physiotherapy for PD and COPD

SUMMARY:
The aim of this study is to investigate whether a smartwatch can measure the physical capacity of patients with Parkinson's Disease and COPD in the physiotherapy practice and at home.

DETAILED DESCRIPTION:
Physical capacity and physical activity are important factors for healthy aging and are found to be predictors of disability, morbidity and mortality in healthy older adults and in people with chronic diseases like Parkinson's Disease and COPD. Physical capacity and activity have mainly been assessed in in-clinic settings using standardized tests and subjective questionnaires. Relying only on in-clinic tests is suboptimal because the tests give limited information on how a patient functions in daily life and cannot capture fluctuations and subtle decrements in disease symptoms. With the rise of innovative technology like wearable sensors, both aspects have become measurable in the patients daily life.

Here, the investigators will study a wrist worn device (The Verily Study Watch) that has the ability to measure physical activity and physical capacity passively and remotely. The primary focus is on its opportunity to measure physical capacity using the 6MWT, referred to as the virtual 6MWT. The watch tags the start and end of the 6 minutes when performing this test. Also, participants can perform the test independently at home. The Study Watch has the options for remote testing of the Timed Up and Go test (TUG) as well. The aim of this study is to investigate whether the virtual 6MWT validly predicts 6MWT outcomes as measured during a supervised, in-clinic test. A valid virtual 6MWT will be extremely valuable for assessing physical capacity in the home situation longitudinally. This will contribute to a more effective and personalized treatment for people with chronic diseases.

The study has a duration of 15 weeks, with 4 in-clinic visits at the physiotherapy practice every five weeks. During those visits, several physical capacity tests will be performed alongside tests and questionnaires related to demographics and disease status. Participants will perform the 6MWT and TUG at home on a weekly basis on a pre-set day and time using the Verily Study Watch. Between week 5 and 15 of the study, participants will follow a standardized aerobic exercise training program according to the most recent regulations.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to read and understand Dutch
* Participant is willing, competent, and able to comply with all aspects of the protocol, including follow-up schedule
* Participant is willing and able to complete patient-reported questionnaires via internet
* Participant can walk
* (PD-specific) Hoehn and Yahr 1-2
* (COPD-specific) Participant has COPD irrespective of airway obstruction severity and has a limited exercise capacity as judged by the physiotherapist

Exclusion Criteria:

* Participant is allergic to nickel
* Participant cannot make an arm swing or is in a situation that prevents arm swing completely
* Co-occurence of COPD and PD
* Participant has cognitive impairment that would prevent understanding and performing tasks in the study
* Participant is pregnant or plans to become pregnant during the course of the study
* Participant is participating in another investigational drug or device study
* Participant has a high fall risk or cardiovascular risk profile
* Participant has any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person with Parkinson's Disease or COPD under treatment or newly referred to the participating physiotherapy practices
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan R Bloem, MD, PhD., Principal Investigator — Radboudumc department of Neurology
Locations (28):
- Netherlands (28):
  - Paca, Aalsmeer
  - Gezondheidscentrum Marne, Amstelveen
  - Fysiotherapie Heusdenhout, Breda
  - Praktijk Graaf Hendrik III Laan, Breda
  - RevaQ, Breda
  - Lijf & leven, fit en fysiotherapie, Ede
  - Fysiotherapie De Hertog, Franeker
  - Zorggroep Ter Weel, Goes
  - Fysio Heerde, Heerde
  - Tigra, Heerenveen
  - Centra Plaza Fysiotherapie, Lelystad
  - Fysiotherapie MTC Lopik, Lopik
  - Vivium Fysiotherapie Naarderheem, Naarden
  - Manueel Fysiocare, Nieuwegein
  - Radboud University Medical Center, Nijmegen
  - FysioHolland Oud Gastel, Oud Gastel
  - Van Broekhoven fysiotherapie, Roosendaal
  - Praktijk Ed van Bruggen, Rotterdam
  - InMotion, Spijkenisse
  - Fysioteam Tegelen, Tegelen
  - Fysiek Vooruit, Teteringen
  - Praktijk Prins Hendrikstraat, The Hague
  - Van der Kieft Fysiotherapie, Uden
  - Motion Fysiotherapie & Preventie, Uithoorn
  - Therapiecentrum Veenstade, Vaassen
  - Fysio van Hoof, expertisecentrum Reva Vitaal, Valkenswaard
  - Rembrandt fysiotherapie & revalidatie, Veenendaal
  - Brabantzorg, Veghel

IPD SHARING:
Plan to Share IPD: Yes
Not decided yet
Supporting Information: Study Protocol, Analytic Code
Time Frame: Not decided yet
Access Criteria: Not decided yet

REFERENCES:
- [Background] de Graaf D, de Vries NM, van de Zande T, Schimmel JJP, Shin S, Kowahl N, Barman P, Kapur R, Marks WJ Jr, van 't Hul A, Bloem BR. Measuring Physical Functioning Using Wearable Sensors in Parkinson Disease and Chronic Obstructive Pulmonary Disease (the Accuracy of Digital Assessment of Performance Trial Study): Protocol for a Prospective Observational Study. JMIR Res Protoc. 2024 May 7;13:e55452. doi: 10.2196/55452. PMID 38713508

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parkinson's Disease | COPD
Started | 89 | 65
Completed | 73 | 56
Not Completed | 16 | 9
Not completed — Withdrawal by Subject | 16 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease | COPD | Total
Number analyzed (Participants) | 89 | 65 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 16 | 48
  >=65 years | 57 | 49 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 59
  Male | 62 | 33 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 89 | 65 | 154
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
6MWT [Mean (Standard Deviation); unit: meter] — Distance walked during the 6MWT
  meter | 413 (92) | 366 (76) | 393 (88)

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Distance Walked During 6MWT
Description: Mean difference in distance walked during the 6MWT (6MWD) derived from the Verily Study Watch and clinician measured distance.
  Note: reported outcome is the mean difference in 6MWD between week 0 and week 15 and is determined as the difference between the two clincian measured distances. The walking distance derived from the Verily Study Watch needs to be determined, this is work in progress
Time Frame: Week 0, week 5, week 10 and week 15
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 89 | 65
meter | 33 (8) | 15 (10)

2. Secondary Outcome: Mean Difference in 6MWD of Study Watch
Description: Difference between 6MWD at home and in-clinic
  Note: not yet reported, data analysis is in progress
Time Frame: Week 0 until week 5
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Change in Physical Capacity
Description: Change in 6MWD from week 5 until week 15 after aerobic exercise capacity training
Time Frame: Week 5 until week 15
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 89 | 65
meters | -17.1 (120.7) | -15.4 (89.1)

4. Secondary Outcome: Mean Difference in TUG Time
Description: Mean difference in time to complete the Timed Up and Go test turing the TUG derived from the verily study watch and clinician measured outcome
  Note: not yet reported, data needs to be analysed
Time Frame: Week 0, Week 5, Week 10, Week 15
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Mean Difference in TUG Time of Study Watch
Description: Difference between TUG time at home and in-clinic
  Note: not yet reported, data needs to be analysed s
Time Frame: Week 0 until week 5
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Change in Gait Speed (10MWT)
Description: The difference in time to complete the 10MWT with and without cognitive task while walking and over time
Time Frame: Week 0, Week 5, Week 10, Week 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 89 | 65
seconds
  Week 0 | -1.3 (2.3) | -1.0 (1.9)
  Week 5 | -1.2 (2.1) | -0.56 (0.6)
  Week 10 | -1.3 (1.9) | -0.4 (0.5)
  Week 15 | -1.2 (1.8) | -0.7 (1.8)

7. Secondary Outcome: Change in Cognition (MoCA)
Description: Change from baseline on the Montreal Cognitive Assessment (MoCA) score at 15 weeks. Range 0-30. Higher scores indicate better cognition
Time Frame: Week 0 and Week 15
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 89 | 65
points
  Week 0 | 25.9 (3.8) | 25.7 (2.7)
  Week 15 | 26.1 (3.8) | 25.2 (2.8)

8. Secondary Outcome: Change in Parkinson's Disease Symptoms (MDS-UPDRS)
Description: Change from baseline in the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) at week 5, week 10 and week 15. Range 0-199. Higher scores indicate worse function.
  note: only the difference in score between week 0 and week 15 is reported
Time Frame: Week 0, Week 5, Week 10, Week 15
Population: COPD participants did not perform this test, as it is a PD-specific test
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 89 | 0
points | 4.5 (19.2) |

9. Secondary Outcome: Change in Self-reported Physical Activity Level (LAPAQ)
Description: Change from baseline on the Longitudinal Aging Study Amsterdam (LASA) physical Activity Questionnaire (LAPAQ)
  Note: not yet reported, data needs to be analysed
Time Frame: Week 0, Week 5, Week 10, Week 15
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Change in Depression and Anxiety (HADS)
Description: Change from baseline on the Hospital Anxiety and Depression Scale (HADS) at week 5, week 10 and week 15. Range 0-42. Higher scores indicate worse function
  Note: only the difference between week 0 and week 15 is reported
Time Frame: Week 0, Week 5, Week 10, Week 15
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 89 | 65
points | 0.6 (3.6) | 0.7 (3.7)

11. Secondary Outcome: Change in Fatigue (FACIT-F13)
Description: Change from baseline on the Functional Assessment of Chronic Illness Therapy (FACIT-F) 13-item at week 5, week 10 and week 15. Range 0-52. Higher scores indicate better function.
  Note: not yet reported, data needs to be analysed
Time Frame: Week 0, Week 5, Week 10, Week 15
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: Change in Sleepiness at Day (ESS)
Description: Change from baseline on the Epworth Sleepiness Scale at week 5, week 10 and week 15. Range 0-24. Higher scores indicate worse function.
  Note: not yet reported, data needs to be analysed
Time Frame: Week 0, Week 5, Week 10, Week 15
Reporting Status: Not Posted, anticipated posting 2025-12

13. Secondary Outcome: Change in Health Related Quality of Life (PDQ-39)
Description: Change from baseline on the Health related quality of life (PDQ-39) questionnaire at week 5, week 10 and week 15. Range 0-100. HIgher scores indicate better function
  Note: only the difference between week 0 and week 15 is reported
Time Frame: Week 0, Week 5, Week 10, Week 15
Population: COPD participants did not complete this questionnaire, as it is a PD-specific questionnaire
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 89 | 0
points | 0.88 (15.3) |

14. Secondary Outcome: Change in Quality of Life (EQ-5D-5L)
Description: Change from baseline in the EQ-5D-5L scores at week 5, week 10 and week 15. Range 0-25. Higher scores indicate worse function
  Note: not yet reported, data data needs to be analysed
Time Frame: Week 0, Week 5, Week 10, Week 15
Reporting Status: Not Posted, anticipated posting 2025-12

15. Secondary Outcome: Clinical COPD Questionnaire (CCQ)
Description: Assessment of and change in health related quality of life from baseline and at week 5, week 10 and week 15. Range 0-60. Higher scores indicate worse function
Time Frame: Week 0, Week 5, Week 10, Week 15
Population: This questionnaire is not completed by the PD participants, as it is an COPD-specific questionnaire
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 0 | 65
score on a scale
  Week 0 |  | 2 [2 to 2]
  Week 5 |  | 2 [1 to 2]
  Week 10 |  | 2 [1 to 2]
  Week 15 |  | 2 [1 to 2]

16. Secondary Outcome: Medical Research Council Dyspnea (mMRC)
Description: Assessment of dyspnea severity at baseline, week 5, week 10 and week 15. Range 0-4. Higher scores indicate worse function
  This test is only completed by the COPD participants as it is a COPD-specific questionnaire.
Time Frame: Week 0, Week 5, Week 10, Week 15
Population: This test is not completed by the PD participants, as it is a COPD-specific questionnaire.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Parkinson's Disease | COPD
Number analyzed (Participants) | 0 | 65
units on a scale
  Week 0 |  | 3 [2 to 3]
  Week 5 |  | 3 [2 to 3]
  Week 10 |  | 3 [2 to 3]
  Week 15 |  | 3 [2 to 3]

17. Secondary Outcome: System Usability Scale (SUS) Questionnaire
Description: Usability of the Verily Study Watch. Range 0-13. Higher scores indicate better usability
Time Frame: Week 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to study completion
Arm/Group | Parkinson's Disease | COPD
All-Cause Mortality (participants affected / at risk) | 0/89 | 1/65
Serious Adverse Events (participants affected / at risk) | 0/89 | 1/65
Other Adverse Events (participants affected / at risk) | 0/89 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson's Disease (N=89) | COPD (N=65)
Lung cancer stage 4 diagnosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT05756075/Prot_SAP_000.pdf